CLINICAL TRIAL: NCT00280631
Title: Phase 1-2a Dose-Ranging Study of TLK199 Tablets in Myelodysplastic Syndrome (MDS)
Brief Title: Study of TLK199 Tablets in Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK199.1101
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2011-06

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — gamma-Glu-S-BzCys-PhGly diethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Dose Escalation Study of TLK199 Tablets From 200 mg Per day To 6000 mg Per Day
  Interventions: Drug: Ezatiostat Hydrochlorine

INTERVENTIONS:
Drug: Ezatiostat Hydrochlorine — Oral Tablets in 2 Divided Doses, Dose Escalation From 200 mg Per Day to 6000 mg Per Day on Days 1-7 of each 21 Day Cycle.
  Other Names: TLK199 Tablets; Telintra

SUMMARY:
The purpose of this study is to determine the safety and efficacy of TLK199 Tablets in patients with Myelodysplastic Syndrome (MDS)

DETAILED DESCRIPTION:
This Phase 1-2a study is an open label, dose-ranging study of TLK199 Tablets in patients with all World Health Organization or French-American-British classification types of myelodysplastic syndrome (MDS). In Phase 1, the safety, pharmacokinetics, and hematologic response rate with TLK199 Tablets will be evaluated. The Phase 1 dose-ranging stage is designed to determine the maximum tolerated dose or optimal biologic dose of TLK199 Tablets. Evaluation of the pharmacokinetics of TLK199 Tablets will be conducted. In Phase 1, an additional 12 patients will undergo pharmacokinetic evaluation under fed conditions at the selected Phase 2a dose. In Phase 2a, further safety and hematologic responses by the modified International Working Group MDS response criteria will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of MDS
* Documented significant cytopenia for at least 2 months
* Adequate liver and kidney function
* Ineligible for stem cell bone marrow transplantation
* At least 18 years of age
* Discontinuation of growth factors (e.g., G-CSF) within 3 weeks of study entry

Exclusion Criteria:

* Prior bone marrow transplant
* Failure to recover from any prior surgery or any major surgery within 4 weeks of study entry
* Pregnant or lactating women
* Other investigational drugs within 14 days of study entry
* Chemotherapy, radiotherapy or immunotherapy within 14 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose or Optimal Biologic Dose | 6 months

SECONDARY OUTCOMES:
Safety Pharmacokinetic Parameters, Hematologic Response Parameters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gail Brown, MD, Study Director — Telik
Locations (3):
- United States (3):
  - Loyola University Chicago-Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Massachusetts (UMass) Memorial Medical Center, Worcester, Massachusetts

REFERENCES:
- [Derived] Raza A, Galili N, Smith S, Godwin J, Lancet J, Melchert M, Jones M, Keck JG, Meng L, Brown GL, List A. Phase 1 multicenter dose-escalation study of ezatiostat hydrochloride (TLK199 tablets), a novel glutathione analog prodrug, in patients with myelodysplastic syndrome. Blood. 2009 Jun 25;113(26):6533-40. doi: 10.1182/blood-2009-01-176032. Epub 2009 Apr 27. PMID 19398716